CLINICAL TRIAL: NCT04924712
Title: Controlled Multicenter Epidemiological Study of Peripheral Leukocyte Populations and Microbiota in Patients With Idiopathic Nephrotic Syndrome (INS)
Brief Title: INS, B Cells and Microbiota
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0118
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Microbiota; B-lymphocytes; Glomerulosclerosis; T-lymphocytes
Keywords: Idiopathic Nephrotic Syndrome; Focal Segmental Glomerulosclerosis; Microbiota; B Lymphocytes; Regulatory T cells
MeSH Terms: conditions — Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with nephrotic syndrome idiopathic: 20 nephrotic INS patients in primary visit: harvesting of 27.5 ml supplementary blood, 40 mlurine and feces at inclusion visit and at 3 months. No intervention, no treatment administration other than usual/routine INS treatment.
  Interventions: Other: Measurement of blood immune populations and microbiota distribution.
- Patient with nephrotic syndrome no idiopathic, IgA or GEM type: 10 NS no idipathic patients: harvesting of 27.5 ml supplementary blood, 40 ml urine and feces at inclusion visit and at 3 months. No intervention, no treatment administration other than usual/routine care treatment.
  Interventions: Other: Measurement of blood immune populations and microbiota distribution.

INTERVENTIONS:
Other: Measurement of blood immune populations and microbiota distribution. — Measurement of peripheral cell populations by spectral cytometry and in parallel, sequencing of intestinal and urinary bacterial 16S RNA of each patient.

SUMMARY:
Idiopathic nephrotic syndrome (NIS) is a clinical entity defined by the association of selective albuminuria, hypoalbuminemia, and nonspecific glomerular lesions (lesions minimal glomerular (LGM) or segmental and focal hyalinosis (HSF). The complication of this kidney disease is the progression towards chronic renal failure and in case of kidney transplantation, its immediate recurrence on the graft . The origin of this syndrome is unknown but a number of clinical observations tend to show an involvement of immune system. A link has been highlighted between atopy, diet and nephrotic flare-ups. The speed of recurrence of this initial disease on the graft and the observation of remissions obtained after treatment by plasma exchange or immunoadsorptions support the presence of a pathogenic plasma factor. Anti-CD20 treatments depleting B lymphocytes has made it possible to favorably treat a number of patients. Dysfunction of regulatory T cells has also been shown in SNI patients. This modification seems linked to allergies and could be due to an aberrant microbiota. The hypothesis of causality between dysbiosis, alteration lymphocyte and triggering of an SNI was mentioned recently. Two studies have shown intestinal dysbiosis in pediatric SNI/LGM, with reduction of T circulating regulators

ELIGIBILITY:
Inclusion Criteria :

* Patient treated in participating centers
* In nephrotic attack, defined biologically by:

Proteinuria > 3g 24h or A proteinuria/creatinuria ratio > 3 or Defined at the discretion of the clinician

Non inclusion Criteria :

* Patient with a history of NIS flare-ups resistant to corticosteroid therapy
* Patient treated with immunosuppressant
* Patient treated with corticosteroids > 10 mg/d
* Weight <50 kg
* Pregnant woman
* Patient under guardianship / curatorship

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with idiopathic nephrotic syndrome (LGM or HSF type) will be considered in the main objective, patients with IgA or GEM type nephrotic syndrome will be integrated into the control group for the secondary objectivets
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2026-01-18 (Estimated); Study Completion 2026-01-18 (Estimated)

PRIMARY OUTCOMES:
Sequencing and analysis of blood peripheral immune populations and intestinal and urinary microbiota | 3 months
  For the analysis of peripheral populations, blood cells will be collected by density gradient (Ficoll) and frozen in 20% DMSO. They will then be marked and identified by flow cytometry.
Sequencing and analysis of intestinal microbiota | 3 months
  The microbiota will be analyzed using DNA extracted from fecal samples.
Sequencing and analysis of urinary microbiota | 3 months
  The microbiota will be analyzed using DNA extracted from urine samples.

SECONDARY OUTCOMES:
Compare blood peripheral immune populations in patients with SNI to that of type SN patients. | 3 months
  We will collect clinical and biological variables from each patient with a syndrome nephrotic type GEM or IgA as well as the results of the analysis of populations peripheral immune systems.
Compare intestinal microbiota in patients with SNI to that of type SN patients. | 3 months
  We will collect clinical and biological variables from each patient with a syndrome nephrotic type GEM or IgA as well as the results of the analysis of the microbiota
Compare urine microbiota in patients with SNI to that of type SN patients. | 3 months
  We will collect clinical and biological variables from each patient with a syndrome nephrotic type GEM or IgA as well as the results of the analysis of the microbiota

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Nantes University Hospital, Nantes, Loire-Atlantique
  - Departemental Hospital Center, La Roche-sur-Yon

IPD SHARING:
Plan to Share IPD: No